CLINICAL TRIAL: NCT03798613
Title: Accuracy of the Apple Watch Series 4 for Detection of Heart Rhythm: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Marc Gillinov, MD, Principal Investigator, The Cleveland Clinic
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 18-1397
Record Dates: First submitted 2018-12-21; First posted 2019-01-10 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Heart Rate Fast; Heart Rate Low
Keywords: Post-op Atrial Fibrillation; Heart Rhythm; Accuracy; Apple Watch
MeSH Terms: conditions — Tachycardia; Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apple Watch 4 Series Device (Active Comparator): Apple watch 4 series heart rate monitoring device
  Interventions: Device: Apple Watch 4 Series Device
- Continuous Telemetry (Active Comparator): Standard continuous telemetry monitoring device
  Interventions: Device: Continuous Telemetry Monitor

INTERVENTIONS:
Device: Apple Watch 4 Series Device — tracings from the apple watch 4 series watch
  Arms: Apple Watch 4 Series Device
Device: Continuous Telemetry Monitor — tracings from the continuous telemetry monitor
  Arms: Continuous Telemetry

SUMMARY:
The objective of this study is to assess the accuracy of the Apple Watch 4 Series watch in generating an ECG that is suitable for determination of heart rhythm compared to rhythms monitored via telemetry. Secondary objective is to assess the accuracy of the Apple Watch 4 series watch in identifying atrial fibrillation when it is present.

DETAILED DESCRIPTION:
The study will assess the accuracy of the Apple watch 4 series watch when worn by post-operative cardiac surgery patients after they have transferred from the ICU to the cardiac telemetry unit.

During testing each subject will wear:

1. An Apple Watch 4 series watch for no more than 5 minutes.
2. Standard continuous telemetry monitor

The location of the watch (left or right wrist) will be randomly assigned.

Heart rate and rhythm will be assessed by obtaining tracings from the Apple Watch 4 series watch while at the same point in time obtaining tracings from a standard telemetry monitor.

ECGs from the Apple Watch 4 will be collected by asking the patient to place his/ her finger on the digital crown of the Apple Watch 4 for 30 seconds. The rhythm displayed by the Apple Watch 4 will be viewed on the Apple health app (available on the iPhone 8) and will be saved for subsequent viewing and analysis.

Each enrolled patient will have a minimum of three assessments of heart rhythm per day for at least two days, generating a minimum of six data points per patient.

After conclusion of the study for each subject, the ECG's from the health app pertaining to that subject will be reviewed by a board certified cardiologist as will the telemetry tracings.

In order to obtain tracings of new onset post-operative atrial fibrillation. 50% of the subjects enrolled will be in sinus rhythm and 50% will be in atrial fibrillation at the time of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Post-operative cardiac surgery patients on the cardiac telemetry floors at the Cleveland Clinic Main Campus

Exclusion Criteria:

* Presence of a cardiac pacemaker
* Use of a radial artery graft for coronary artery bypass grafting
* Tattoos located on the skin of the wrist or forearm where the Apple Watch 4 will be placed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Heart rate accuracy compared to telemetry | 5 minutes
  Apple Watch 4 Series heart rate monitor device accuracy compared to standard continuous telemetry monitor. This will be expressed by the correlation coefficient.

SECONDARY OUTCOMES:
Heart rhythm accuracy compared to telemetry | 5 minutes
  Apple Watch 4 Series heart rhythm device accuracy compared to standard continuous telemetry monitor. This will be expressed by the correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Gillinov, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States